CLINICAL TRIAL: NCT03442166
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial on the Effectiveness of Light-emitting Diode (LED) Photobiomodulation in Pain Management, Facial Edema, Trismus and Quality of Life After Extraction of Retained Lower Third Molars
Brief Title: Effectiveness of Light-emitting Diode (LED) Photobiomodulation in the Extraction of Retained Lower Third Molars
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Carlos
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Pain, Postoperative; Edema; Trismus; Quality of Life
MeSH Terms: conditions — Pain, Postoperative; Edema; Trismus

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: After the suture is completed, the researcher responsible for applying the LED will remove and open the envelope containing the information from the experimental group in which the patient will be inserted and proceed to the experiment. A single examiner will run the daily application of the LED and will not perform any type of evaluation. Surgical procedures will be performed by the same surgeon. The preoperative and postoperative evaluations (1, 2, 5 and 7 days postoperatively) will be done by an examiner who will not be aware of the group in which each patient is allocated. Patients will not be aware of whether or not they received LED irradiation, because the person in charge of the LED application will position the plate in place for intra and extraoral irradiation in all patients and only trigger the light when and where predicted in the specific experimental group. The characteristic sound of the device will be triggered by recording in the sham group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LED group (Active Comparator): The patients (n=17) will receive daily intra and extra oral LED applications from the immediate postoperative period up to 7 days after the surgical procedure. The LED irradiation will be performed in two areas, one intra and one extra oral. The LED to be used in the intraoral site will be red, 660+/-20nm wavelength, 5 mW power, 2.7J/cm2 energy density for 7 min, 2J energy per point, knowing that the 6 irradiated spots will have 12J in total. In the extra oral site the infra-red LED will be used, 850+/-20nm wavelength, power of 5mW, 3.8J/cm2 of energy density for 10 min, 3J of energy per point, knowing that 36 will be irradiated, so we will have 108J in total.
  Interventions: Radiation: LED group
- Sham group (Sham Comparator): Patients (n=17) will be treated in the same way as the LED group. The person in charge of the application will simulate the intraoral and extraoral irradiation by positioning the LED in the same locations described for the LED group, but the equipment will be kept off. So that the patient does not identify the sound of activation of the device (beep), it will be recorded, and connected at the time of application.
  Interventions: Radiation: Sham group

INTERVENTIONS:
Radiation: LED group — The patients (n=17) will receive daily intra and extra oral LED applications from the immediate postoperative period up to 7 days after the surgical procedure. The LED irradiation will be performed in two areas, one intra and one extra oral. The LED to be used in the intraoral site will be red, 660+/-20nm wavelength, 5 mW power, 2.7J/cm2 energy density for 7 min, 2J energy per point, knowing that the 6 irradiated spots will have 12J in total. In the extra oral site the infra-red LED will be used, 850+/-20nm wavelength, power of 5mW, 3.8J/cm2 of energy density for 10 min, 3J of energy per point, knowing that 36 will be irradiated, so we will have 108J in total.
  Arms: LED group
Radiation: Sham group — Patients will be treated in the same way as the LED group. The person in charge of the application will simulate the intraoral and extraoral irradiation by positioning the LED in the same locations described for the LED group, but the equipment will be kept off. So that the patient does not identify the sound of activation of the device (beep), it will be recorded, and connected at the time of application.
  Arms: Sham group

SUMMARY:
In dentistry, one of the most common surgical procedures is the removal of included third molars. This surgery generates great morbidity to patients for causing pain, edema and trismus due to surgical trauma. The use of photobiomodulation (PBM) (low-power laser or light emitting diode - LED) in the postoperative of these procedures has shown excellent results in the control of postoperative sequelae. The objective of the present study is to evaluate the effectiveness of PBM with LED in the control of pain, facial edema, trismus and quality of life resulting from the extraction of retained lower third molars. A randomized, double-blind, placebo-controlled clinical trial involving 34 adult patients, who search the Discipline of Buccomaxillofacial Surgery and Traumatology (CTBMF) II of FO-UFRGS for the removal of included lower third molars will be conducted. Before and after the surgeries, the facial and mouth opening measurements of all patients will be done. Immediately after the surgeries, the patients will be randomized by means of envelopes in two groups. In the LED group the patients will receive daily LED applications (intra oral with 660nm and extra oral with 850nm) from the immediate postoperative to 7 days after the surgical procedure. In the control group the patients will be treated in the same way as in the LED group, however, the person in charge of the application will simulate intraoral and extraoral irradiation with the LED kept off. Pain (EVA and NRS-101), postoperative edema, trismus, temperature, dysphagia and hematomas, as well as the impact of the surgical procedure on patients' quality of life will be evaluated after 1, 2, 5 and 7 days. For the analysis of the oral health impact profile (OHIP-14 Questionnaire) and anxiety analysis (Beck anxiety inventory -BAI) the questionnaires will be applied preoperatively and 7 days after treatment. Initial descriptive analyzes will be performed considering all variables measured in the study, both quantitative (mean and standard deviation) and qualitative (frequencies and percentages). Later, the appropriate statistical tests will be applied for each specific analysis. In all tests, the significance level of 5% probability or the corresponding p-value will be adopted. All analyzes will be performed using the statistical software SAS for Windows, version 9.1.3.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need surgical removal of retained lower third molars;
* Patients who agree to participate in the study after reading and signing the Term of Consent for Participation in Clinical Research.
* Patients with indication for extraction of lower third molars (recurrent infections, bad position, orthodontic indication) or written professional indication (ASA I - negative medical history), systolic blood pressure less than 140mmHg, and diastolic blood pressure lower than 90mmHg and heart rate values of 70 ± 20 beats / minute and have the upper and lower central incisor teeth.

Exclusion Criteria:

* Patients who have systemic diseases, chronic pain or neurological and psychiatric disorders;
* Claim to be smokers;
* Are using anti-inflammatories, analgesics or bisphosphonates in the last 15 days;
* Present active pericoronaritis;
* Are pregnant;
* are breastfeeding;
* Severe temporomandibular disorders
* Have photo sensitivity history
* Are allergic to any drug used in the research (paracetamol, chlorhexidine 2%)
* Patients presenting radiolucent images associated with the teeth to be extracted
* Patients who present any type of complication during surgery (hemorrhage, operative difficulty, time greater than 90 minutes of surgery), as these cases are not in the standard expected for third molar surgeries. In this case the central action analgesic will be prescribed. These data will not be part of the statistical analysis but will be described and discussed as well as possible adverse effects.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in postoperative pain | After 1, 2, 5 and 7 days of surgeries.
  A Visual Analog Scale (VAS) will be printed on the patient evaluation form and the subjects will be instructed by the evaluator to mark a point in the line of 10 cm, indicating the intensity of their pain after 1,2, 5 and 7 days of the surgeries.

SECONDARY OUTCOMES:
Changes of postoperative edema | After 1, 2, 5 and 7 days of surgeries.
  The evaluator will measure the distances between the corner of the eye and angle of the mandible, between the tragus and labial commissure and between the tragus and pogonium.
Change of trismus | After 1, 2, 5 and 7 days of surgeries.
  The evaluator will measure the opening of the mouth using a pachymeter in each patient 1, 2, 5 and 7 days after surgery.
Changes in quality of life | Before and 7 days after surgery.
  The Oral Health Impact Profile (OHIP-14) is a simplified form of the original OHIP questionnaire that is used to assess the impact of oral health on subjects' quality of life. The items are distributed among the following subscales: functional limitation, pain, psychological discomfort, physical disability, psychological deficiency, social incapacity and disability. The questionnaire will be applied by the evaluator.
Changes in postoperative pain (NRS-10 scale) | After 1, 2, 5 and 7 days of surgeries.
  For the NRS-101 scale, the evaluators will ask patients to assign a number between 0 (no pain) and 100 (worst possible pain) that best represents the pain they are currently experiencing after 1, 2, 5 and 7 days of surgeries.

CONTACTS AND LOCATIONS:
Locations (1):
- UniNove, São Paulo, São Paulo, Brazil